CLINICAL TRIAL: NCT00437554
Title: A 16-Week Controlled, Double Blind, Double Dummy, Randomized, Two Arm Parallel-Group Study to Compare the Efficacy and Safety of Amaryl M 1/250 mg b.i.d vs. Amaryl M SR 2/500 mg od. in Patients With Type 2 Diabetes Mellitus
Brief Title: Phase III Study for Glimepiride + Metformin Hydrochloride (Amaryl M) Slow Release (SR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLIME_L_01019
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Glimepiride

SUMMARY:
Primary:

To show the equivalence in terms of efficacy glycated hemoglobin (HbA1c) of glimepiride/metformin slow-release combination tablet (Amaryl M SR 2/500) once daily compared with fixed-dose glimepiride/metformin combination tablet (Amaryl M 1/250) twice a day on HbA1c in patients with type 2 Diabetes Mellitus (DM)

Secondary: To compare the following parameters in two treatment arm

* Efficacy; Fasting Plasma Glucose (FPG) and Post-prandial two hours plasma glucose (PP2h)
* Response rates in terms of HbA1c, FPG
* Patient compliance

Safety:

* episodes of hypoglycemia
* adverse events
* laboratory values including hematology blood chemistry and urinalysis
* vital sign and physical examination

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 DM diagnosed for at least 3 months but no longer than 10 years before screening;
* - BMI ≤ 40 kg/m²;
* A negative pregnancy test for all females of childbearing potential

Exclusion Criteria:

* A history of acute metabolic complications such as diabetic ketoacidosis or hyperosmolar nonketotic coma within 3 months before screening;
* Current therapy with any oral anti-diabetic drugs or previous use in the 4 weeks other than sulfonylureas or metformin (8 weeks in case of thiazolidinedione) before screening;
* Concomitant treatment prohibited during the study period;
* Any oral anti-diabetic drugs other than study medication
* Any insulin therapy over 7 days consecutively or intermittently in order to treat acute metabolic decompensation or systemic infection during the study
* Intermittent use of systemic corticosteroids or large dose of inhaled steroids
* Subjects with clinically significant renal (serum creatinine level >1.5 mg/dL in male and >1.4 mg/dL in female) or hepatic disease (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2x upper limit of normal (ULN));
* Subjects with acute and severe cardiovascular disease (e.g. heart failure, myocardiac infarction, stroke etc.)
* Clinically significant laboratory abnormality on screening labs or any medical condition that would affect the completion or outcome of the study in the opinion of the investigator and/or sponsor;
* Pregnant or lactating females;
* History of drug or alcohol abuse;
* Subjects with known hypersensitivity to glimepirides, or metformin; Night-shift workers;
* Treatment with any investigational product in the last 3 months before study entry;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2006-08; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Efficacy : Change in HbA1c between baseline and endpoint

SECONDARY OUTCOMES:
Efficacy : Change in HbA1c measured at baseline, week 8 and week 16. Change in FPG and PP2h measured at baseline, week 8 and week 16. Response rates in terms of HbA1c, FPG.Patient compliance
Safety: episodes of hypoglycemia, adverse events, laboratory values including hematology, blood chemistry and urinalysis, vital sign and physical examination, Frequency with hypoglycemic episode

CONTACTS AND LOCATIONS:
Overall Officials: Hyou-Young Rhim, Study Director — Handok Inc.
Locations (1):
- Handok, Seoul, South Korea